CLINICAL TRIAL: NCT04805619
Title: Evaluation of the Neointimal Healing by OCT of the Tapered DES Biomime Morph (TAPER-I Study)
Acronym: TAPER-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Henrique Barbosa Ribeiro, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Instituto do Coração
Record Dates: First submitted 2021-03-12; First posted 2021-03-18 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Stent; Long coronary lesions; Angioplasty; Neointimal healing; Tapering
MeSH Terms: conditions — Atherosclerosis | interventions — Stents

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open-label study, including patients presenting at least one long or very long lesion (≥ 30 mm), who will undergo angioplasty with a tapered DES
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients with long or very long lesions (≥ 30 mm) in native coronary arteries.
  Interventions: Device: Biomime Morph, a tapered drug eluting stent (DES) with hybrid design

INTERVENTIONS:
Device: Biomime Morph, a tapered drug eluting stent (DES) with hybrid design — Biomime Morph DES is a cobalt-chromium stent, with strut thickness of 65 µm, a hybrid cell design (closed cells in the extremity and open cells in the middle) and a conic shape, where the proximal part of the stent is 0.5 mm larger than the distal part (Table 1). In addition, the Biomime Morph elutes Sirolimus from a biodegradable polymer matrix.
  Other Names: Stent

SUMMARY:
The long and very long stents, although they represent a greater navigability challenge, especially in tortuous and calcified coronary arteries, they have the advantage of providing shorter procedural time, with less contrast use, less exposure to radiation, lower cost, lower risk of occlusion of lateral branches, as well as less interference in the local flow. However, in the context of the use of such long stents, as some vessels have a tapering shape, with a progressively smaller diameter in their more distal segments (as is the typical case of the left anterior descending artery), a significant disproportion (mismatch) of vessel size between the proximal and distal landing zone of the stent can be noted. Such disproportion may lead to the underestimation of the proximal reference or overestimation of the distal reference diameter of the vessel, generating an increase of the stress on the vessel wall, with consequent increase in the risk of restenosis. In view of this situation, long or very long stents were developed in a tapered shape, with progressive reduction of their diameter between their proximal and distal portion, respecting the phenomenon of tapering of the coronary artery during the treatment of very long lesions.Some of these stents also have a hybrid design, with closed cells at the ends and open cells in the middle, allowing a more efficient expansion in their middle portion (thus avoiding the dog-boning phenomenon). However, there is still a lack of studies in the literature evaluating whether these DES in a tapered shape and hybrid cells may effectively heal over time, specially with respect to strut covering and strut malapposition. Thus, this is a prospective, single-arm, open-label study, including patients presenting at least one long or very long lesion (≥ 30 mm), who will undergo angioplasty with a tapered DES. The objective is to analyze the neointimal healing as well as other data on the efficacy and safety of the tapered DES Biomime Morph in patients with long or very long lesions.

ELIGIBILITY:
Inclusion Criteria:

* General clinical criteria

  * Both gender with age ≥ 18 years
  * Clinical indication for a PCI with a DES due to an acute coronary syndrome for unstable angina or non-ST elevation myocardial infarction (NSTEMI), stable angina, or in asymptomatic patients with objective evidence of ischemia.
  * Included patients must have all inclusion criteria and provide written informed consent.
* Angiographic criteria

  * Lesions with a length ≥ 30 mm, amenable for the treatment with only one stent
  * Up to 2 "de novo" lesions/patients in native vessels
  * Vessel diameter between 2.5 and 4 mm.

Exclusion Criteria:

* General clinical exclusion criteria

  * Previous use of brachytherapy or a stent in the target vessel;
  * Left ventricular ejection fraction <25%;
  * bleeding diathesis;
  * Contraindication to aspirin or P2Y12 inhibitors, heparina or any component of the DES.
  * Creatinine levels > 2.0mg/dl;
  * Leucocyte count < 3.500 céls/mm3;
  * Platelet count < 100.000 céls/mm³
  * Pregnancy;
  * Surgical procedure scheduled within the next 6 months, except if DAPT could be maintained;
  * Impossibility to provide written informed consent.
* Angiographic Criteria

  * Left main disease > 50%;
  * Bifurcation lesions with side branch > 2.0mm in diameter where a stent should be required in the side branch (2-stent technique);
  * Occluded vessel (Thrombolysis in Myocardial Infaction grade 0 /1)
  * Restenosis;
  * Saphenous vein graft and LIMA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the stent coverage and neo-intimal growth assessed at six months. The neointimal healing score is based on four scaffold- or stent-related characteristics and is calculated on a lesion level: | Six months
  1. Presence of filling defect (% intraluminal defect, ILD) is assigned a weight of "4"
  2. Presence of both malapposed and uncovered struts (% malapposed/uncovered, MU) is assigned a weight of "3"
  3. Presence of uncovered struts alone (% malapposed, M) is assigned a weight of "2"
  4. Presence of malapposed struts alone (% uncovered, U) is assigned a weight of "1" Neointimal healing score = (%ILD * 4)+(%MU * 3)+(%U * 2)+(%M * 1).

SECONDARY OUTCOMES:
Major adverse cardiac events and Stent Thrombosis | 30 days, 6 months and 1 year
  * Major adverse cardiac events (MACE), defined as a composite of death, nonfatal myocardial infarct or target vessel revascularization, at 30 days, 6 months and 1 year.
  * Stent thrombosis at 1 year.
Efficacy secondary endpoints | 6 months and 12 months
  * Angiographic success
  * Procedure success
  * Target lesion revascularization (TLR) at 6 and 12 months
  * Target vessel revascularization (TVR) at 6 and 12 months
  * Modified neointimal healing score, calculated at 6 months
  * Intra-segment luminal loss (intra-stent segment and proximal and distal 5 mm edges) at 6 months
  * Intra-stent luminal loss at 6 months
  * Intra-stent and intra-segment binary restenosis
  * Percentage of neointimal obstruction
  * Intra-stent mean percentage neointimal obstruction by the optical frequency domain image (OFDI)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coração - HCFMUSP, São Paulo, Brazil

REFERENCES:
- [Background] Berry D. The unlocking of the coronary arteries: origins of angioplasty. A short historical review of arterial dilatation from Dotter to the creative Gruentzig. Eur Heart J. 2009 Jun;30(12):1421-2. doi: 10.1093/eurheartj/ehp182. No abstract available. PMID 19525552
- [Background] Honda Y, Muramatsu T, Ito Y, Sakai T, Hirano K, Yamawaki M, Araki M, Kobayashi N, Takimura H, Sakamoto Y, Mouri S, Tsutumi M, Takama T, Takafuji H, Tokuda T, Makino K. Impact of ultra-long second-generation drug-eluting stent implantation. Catheter Cardiovasc Interv. 2016 Feb 1;87(2):E44-53. doi: 10.1002/ccd.26010. Epub 2015 May 23. PMID 26010548
- [Background] Bouras G, Jhamnani S, Ng VG, Haimi I, Mao V, Deible R, Cao S, Sudhir K, Lansky AJ. Clinical outcomes after PCI treatment of very long lesions with the XIENCE V everolimus eluting stent; Pooled analysis from the SPIRIT and XIENCE V USA prospective multicenter trials. Catheter Cardiovasc Interv. 2017 May;89(6):984-991. doi: 10.1002/ccd.26711. Epub 2016 Aug 22. PMID 27545721
- [Background] Sgueglia GA, Belloni F, Summaria F, Conte M, Cortese B, Silva PL, Ricci R, Lioy E, Pucci E, Gaspardone A. One-year follow-up of patients treated with new-generation polymer-based 38 mm everolimus-eluting stent: the P38 study. Catheter Cardiovasc Interv. 2015 Feb 1;85(2):218-24. doi: 10.1002/ccd.25542. Epub 2014 May 26. PMID 24824088
- [Background] Meier B, Gruentzig AR, Hollman J, Ischinger T, Bradford JM. Does length or eccentricity of coronary stenoses influence the outcome of transluminal dilatation? Circulation. 1983 Mar;67(3):497-9. doi: 10.1161/01.cir.67.3.497. PMID 6217920
- [Background] Kornowski R, Bhargava B, Fuchs S, Lansky AJ, Satler LF, Pichard AD, Hong MK, Kent KM, Mehran R, Stone GW, Leon MB. Procedural results and late clinical outcomes after percutaneous interventions using long (> or = 25 mm) versus short (< 20 mm) stents. J Am Coll Cardiol. 2000 Mar 1;35(3):612-8. doi: 10.1016/s0735-1097(99)00580-x. PMID 10716462
- [Background] Schalij MJ, Udayachalerm W, Oemrawsingh P, Jukema JW, Reiber JH, Bruschke AV. Stenting of long coronary artery lesions: initial angiographic results and 6-month clinical outcome of the micro stent II-XL. Catheter Cardiovasc Interv. 1999 Sep;48(1):105-12. doi: 10.1002/(sici)1522-726x(199909)48:13.0.co;2-0. PMID 10467083
- [Background] Kobayashi Y, De Gregorio J, Kobayashi N, Akiyama T, Reimers B, Finci L, Di Mario C, Colombo A. Stented segment length as an independent predictor of restenosis. J Am Coll Cardiol. 1999 Sep;34(3):651-9. doi: 10.1016/s0735-1097(99)00303-4. PMID 10483943
- [Background] Kobayashi Y, De Gregorio J, Kobayashi N, Reimers B, Albiero R, Vaghetti M, Finci L, Di Mario C, Colombo A. Comparison of immediate and follow-up results of the short and long NIR stent with the Palmaz-Schatz stent. Am J Cardiol. 1999 Sep 1;84(5):499-504. doi: 10.1016/s0002-9149(99)00366-5. PMID 10482144
- [Background] Di Sciascio G, Patti G, Nasso G, Manzoli A, D'Ambrosio A, Abbate A. Early and long-term results of stenting of diffuse coronary artery disease. Am J Cardiol. 2000 Dec 1;86(11):1166-70. doi: 10.1016/s0002-9149(00)01197-8. PMID 11090785
- [Background] Kastrati A, Elezi S, Dirschinger J, Hadamitzky M, Neumann FJ, Schomig A. Influence of lesion length on restenosis after coronary stent placement. Am J Cardiol. 1999 Jun 15;83(12):1617-22. doi: 10.1016/s0002-9149(99)00165-4. PMID 10392864
- [Background] Saucedo JF, Kennard ED, Popma JJ, Talley D, Lansky A, Leon MB, Baim DS. Importance of lesion length on new device angioplasty of native coronary arteries. NACI Investigators. New Approaches to Coronary Interventions. Catheter Cardiovasc Interv. 2000 May;50(1):19-25. doi: 10.1002/(sici)1522-726x(200005)50:13.0.co;2-h. PMID 10816274
- [Background] Kornowski R, Mehran R, Hong MK, Satler LF, Pichard AD, Kent KM, Mintz GS, Waksman R, Laird JR, Lansky AJ, Bucher TA, Popma JJ, Leon MB. Procedural results and late clinical outcomes after placement of three or more stents in single coronary lesions. Circulation. 1998 Apr 14;97(14):1355-61. doi: 10.1161/01.cir.97.14.1355. PMID 9577946
- [Background] Applegate RJ, Sacrinty MT, Kutcher MA, Santos RM, Gandhi SK, Little WC. Effect of length and diameter of drug-eluting stents versus bare-metal stents on late outcomes. Circ Cardiovasc Interv. 2009 Feb;2(1):35-42. doi: 10.1161/CIRCINTERVENTIONS.108.805630. Epub 2009 Feb 10. PMID 20031691
- [Background] Shirai S, Kimura T, Nobuyoshi M, Morimoto T, Ando K, Soga Y, Yamaji K, Kondo K, Sakai K, Arita T, Goya M, Iwabuchi M, Yokoi H, Nosaka H, Mitsudo K; j-Cypher Registry Investigators. Impact of multiple and long sirolimus-eluting stent implantation on 3-year clinical outcomes in the j-Cypher Registry. JACC Cardiovasc Interv. 2010 Feb;3(2):180-8. doi: 10.1016/j.jcin.2009.11.009. PMID 20170875
- [Background] Degertekin M, Arampatzis CA, Lemos PA, Saia F, Hoye A, Daemen J, Tanabe K, Lee CH, Hofma SJ, Sianos G, McFadden E, van der Giessen W, Smits PC, de Feyter PJ, van Domburg RT, Serruys PW. Very long sirolimus-eluting stent implantation for de novo coronary lesions. Am J Cardiol. 2004 Apr 1;93(7):826-9. doi: 10.1016/j.amjcard.2003.12.018. PMID 15050483
- [Background] Lee CW, Park DW, Lee BK, Kim YH, Hong MK, Kim JJ, Park SW, Park SJ. Predictors of restenosis after placement of drug-eluting stents in one or more coronary arteries. Am J Cardiol. 2006 Feb 15;97(4):506-11. doi: 10.1016/j.amjcard.2005.09.084. Epub 2006 Jan 4. PMID 16461047
- [Background] Kastrati A, Dibra A, Mehilli J, Mayer S, Pinieck S, Pache J, Dirschinger J, Schomig A. Predictive factors of restenosis after coronary implantation of sirolimus- or paclitaxel-eluting stents. Circulation. 2006 May 16;113(19):2293-300. doi: 10.1161/CIRCULATIONAHA.105.601823. Epub 2006 May 8. PMID 16682614
- [Background] Tsagalou E, Chieffo A, Iakovou I, Ge L, Sangiorgi GM, Corvaja N, Airoldi F, Montorfano M, Michev I, Colombo A. Multiple overlapping drug-eluting stents to treat diffuse disease of the left anterior descending coronary artery. J Am Coll Cardiol. 2005 May 17;45(10):1570-3. doi: 10.1016/j.jacc.2005.01.049. PMID 15893168
- [Background] Hoffmann R, Herrmann G, Silber S, Braun P, Werner GS, Hennen B, Rupprecht H, vom Dahl J, Hanrath P; IMPact Upon Long Lesion StEnting Study Group. Randomized comparison of success and adverse event rates and cost effectiveness of one long versus two short stents for treatment of long coronary narrowings. Am J Cardiol. 2002 Sep 1;90(5):460-4. doi: 10.1016/s0002-9149(02)02514-6. PMID 12208402
- [Background] Timmins LH, Meyer CA, Moreno MR, Moore JE Jr. Mechanical modeling of stents deployed in tapered arteries. Ann Biomed Eng. 2008 Dec;36(12):2042-50. doi: 10.1007/s10439-008-9582-0. Epub 2008 Oct 10. PMID 18846425
- [Background] Hehrlein C, DeVries JJ, Arab A, Haller SD, Kloostra A, Lauer MA, Foster MT, Fischell TA. Role of the "dogbone" effect of balloon-expandable stents: quantitative coronary analysis of DUET and NIR stent implantation introducing a novel indexing system. J Invasive Cardiol. 2002 Feb;14(2):59-65. PMID 11818639
- [Background] Valero E, Consuegra-Sanchez L, Minana G, Garcia-Blas S, Rodriguez JC, Moyano P, Sanchis J, Nunez J. Initial experience with the novel BioMime 60 mm-long sirolimus-eluting tapered stent system in long coronary lesions. EuroIntervention. 2018 Jan 20;13(13):1591-1594. doi: 10.4244/EIJ-D-17-00616. No abstract available. PMID 28870879
- [Background] Premchand RK, Kumar YS. A Report of Successful Procedural, Clinical, and Angiographic Outcomes with a Tapered Stent of a Patient in Naturally Tapered Coronary Vessel. J Clin Diagn Res. 2017 Jan;11(1):OD06-OD07. doi: 10.7860/JCDR/2017/22241.9288. Epub 2017 Jan 1. PMID 28273994
- [Background] Menown IB. Very long stent technology: clinical and practical value. Future Cardiol. 2013 Sep;9(5):641-4. doi: 10.2217/fca.13.50. No abstract available. PMID 24020665
- [Background] Raber L, Onuma Y, Brugaletta S, Garcia-Garcia HM, Backx B, Iniguez A, Okkels Jensen L, Cequier-Fillat A, Pilgrim T, Christiansen EH, Hofma SH, Suttorp M, Serruys PW, Sabate M, Windecker S. Arterial healing following primary PCI using the Absorb everolimus-eluting bioresorbable vascular scaffold (Absorb BVS) versus the durable polymer everolimus-eluting metallic stent (XIENCE) in patients with acute ST-elevation myocardial infarction: rationale and design of the randomised TROFI II study. EuroIntervention. 2016 Jul 20;12(4):482-9. doi: 10.4244/EIJY15M08_03. PMID 26342471